CLINICAL TRIAL: NCT05361317
Title: Correction of Hallux Valgus with the Nexis® PECA Bunion Implantable Osteosynthesis Medical Device : Evaluation of Quality of Life Scores, Angular Correction, Bone Consolidation and Occurrence of Adverse Events
Brief Title: Correction of Hallux Valgus with the Nexis® PECA Bunion Implantable Osteosynthesis Medical Device
Acronym: PECA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novastep (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-1
Record Dates: First submitted 2022-04-22; First posted 2022-05-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-06

CONDITIONS: Hallux Valgus
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hallux valgus correction (Other): Hallux valgus correction for all patients : intervention during intraoperative visit, with Nexis® PECA Bunion Implantable Osteosynthesis Medical Device
  Interventions: Device: Nexis® PECA Bunion device

INTERVENTIONS:
Device: Nexis® PECA Bunion device — Hallux valgus correction with percutaneous chevron and Akin osteotomy.

SUMMARY:
The Nexis® screw system is a range of osteosynthesis screws for the foot. Nexis® Bunion Screws are Class IIb implantable medical devices.

The primary objective of the study is to confirm the performance and effectiveness of the device under investigation for the correction of hallux valgus with the evaluation functional capacities of the patient's foot. It will be assessed with "general sub-score" of the EFAS questionnaire determined during the postoperative visit at 6 months.

The evaluation of quality of life scores, angular correction, bone consolidation and occurrence of adverse events will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a hallux valgus foot pathology requiring correction
* First line operation
* Use of the medical device concerned PECA Bunion
* Unilateral operation
* Patient aged 18 or over
* Isolated hallux valgus correction, without associated surgical procedures
* Patient able to respect the prescriptions and recommendations of his surgeon
* Patient able to read and understand the information note on the objectives of the study and the collection of their data
* Patient able to sign a consent form

Exclusion Criteria:

* Patient with a contraindication to the device under investigation,
* Simultaneous participation in another clinical investigation protocol,
* Adults subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty, pregnant or breastfeeding women, minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2026-06-13 (Estimated)

PRIMARY OUTCOMES:
Confirm performance and effectiveness of the device under investigation for the correction of hallux valgus in terms of functional capacities of patient's foot determined thanks to the "general sub-score" of the European Foot and Ankle Society scale | 6 months post-operative
  Confirm the performance and effectiveness of the device under investigation for the correction of hallux valgus in terms of functional capacities of the patient's foot, with the evaluation of the "general sub-score" of the European Foot and Ankle Society (EFAS) questionnaire during post-operative visit at 6 months.
  The questionnaire collects information on the following categories: functional capacity of the patient's foot in general (6 items), and functional capacity of the patient's foot during sport (4 items).
  The scores to be calculated range from 0-4 per question, 0-24 for the general category (the only category to be evaluated for the primary outcome).
  A score of 0 indicates the worst possible foot/ankle symptoms and 24 indicates no symptoms foot/ankle.
  In this study, an objective score of 16 (out of a total of 24) was determined

SECONDARY OUTCOMES:
Confirm performance and effectiveness of the device under investigation for the correction of hallux valgus with the evaluation of clinical parameters with the evaluation of the evolution of the pain with Visual Analog Scale | 6-8 weeks, 3-4 months, 6 months and 2 years post-operative
  The VAS (Visual Analog Scale) score is a tool used to measure pain ranging from 0 (no pain) to 10 (very intense pain).
  An evolution of 4.63 is expected between preoperative visit and postoperative visits
Confirm performance and effectiveness of the device under investigation for the correction of hallux valgus with evaluation of clinical parameters: evaluation of the evolution of the quality of life with American Orthopedic Foot and Ankle Scale | 3-4 months, 6 months and 2 years post-operative
  The American Orthopedic Foot and Ankle Score (AOFAS) combines subjective pain and function scores provided by the patient and objective scores based on the physician's physical examination. The questionnaire is composed of nine items, divided into three categories: pain, functional aspects and alignment, resulting in a total score of 100 points. A score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  An improvement of 26.87 in the AOFAS score is expected at postoperative visits compared to preoperative visit.
Confirm the performance and effectiveness of the device under investigation for the correction of hallux valgus with the evaluation of clinical parameters : evaluation of the evolution of the quality of life with The Short Form (36) Health Survey | 6 months and 2 years post-operative
  The Short Form (36) Health Survey is a standardized auto-questionnaire for measuring quality of life. The questionnaire is made up of 36 questions, divided into 8 dimensions: physical activity, life and relationships with others, physical pain, perceived general health, vitality, limitations due to mental state, limitations due to physical state, mental health.
  SF-36 is a 0-100 scale : a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  An improvement of 3.6 in the SF-36 score is expected at postoperative visits compared to preoperative visit
Confirm performance and effectiveness of the device for the correction of hallux valgus with the evaluation of clinical parameters: evaluation of functionality of the foot in sport with "sub-score sport" of the European Foot and Ankle Society scale | 3-4 months, 6 months and 2 years post-operative
  The sport sub-score of the European Foot and Ankle Society (EFAS) questionnaire is used to measure the functional capacity of the patient's foot during sports practice and ranges from 0 to 16 for the sport category, with a score of 0 indicating the worst possible foot/ankle symptoms and 16 indicating no foot/ankle symptoms.
  An improvement of 4.7 in the sub-score "sport" of the EFAS is expected at postoperative visits
Confirm performance and effectiveness of the device for the correction of hallux valgus with the evaluation of radiographics parameters: evaluation of evolution of angular measures (hallux valgus, Inter-metatarsal and Distal Metaphyseal Articular Angles) | 6-8 weeks, 3-4 months, 6 months and 2 years post-operative
  Hallux valgus angle (HVA), Inter-metatarsal angle (IMA) and Distal Metaphyseal Articular Angle (DMAA) are calculated with radiography.
  The expected angle correction is a reduction of 7.60° for HVA, 4° for IMA and 5.50° for DMAA at 6 months and 2 years postoperative.
Confirm the performance and effectiveness of the device under investigation for the correction of hallux valgus with the evaluation of radiographics parameters (X-rays) with the evaluation of evolution of consolidation | 6-8 weeks, 3-4 months, 6 months and 2 years post-operative
  The evaluation of bone consolidation on x-rays will be carried out by the surgeon. The presence of bone consolidation at a rate greater than or equal to 90% should be demonstrated at 6-8 weeks, 3-4 months, 6 months and 2 years postoperatively.
Confirm the performance and effectiveness of the device under investigation for the correction of hallux valgus with the evaluation of clinical parameters thanks to the evaluation of mobility (dorsiflexion and plantar flexion) | 6-8 weeks, 3-4 months, 6 months and 2 years post-operative
  Description and comparison of:
  Dorsiflexion mobility at V2 (6-8 weeks), V3 (3-4 months), 6 months (V4) and at 2 years (V5) compared to V0 : A mobility greater than or equal to 57.35° is expected.
  and Mobility in plantar flexion at V2 (6-8 weeks), V3 (3-4 months), 6 months (V4) and at 2 years (V5) compared to V0 : A mobility of 24.85° is expected.
Confirm the safety of the device under investigation for the correction of hallux valgus by evaluating the occurrence of adverse events, complications and device defects | From inclusion visit (V0) to 2 years post-operative visit
  The occurrence of adverse events (including complications) and defects will be assessed intraoperatively and at each postoperative visit by questioning the patient, clinical and radiographic examinations.

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Girod, Study Director — Novastep
Locations (4):
- France (4):
  - New Clinic Bel Air, Bordeaux
  - Policlinic Bordeaux North Aquitaine, Bordeaux
  - Saint-Charles Clinic, Lyon
  - Toulouse University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided